CLINICAL TRIAL: NCT05173805
Title: Phase I Clinical Study on the Safety, Tolerance, Pharmacokinetics and Efficacy of YL-15293 in Patients With Advanced Solid Tumor With KRAS Mutation
Brief Title: Phase I Clinical Study of YL-15293 in Patients With Advanced Solid Tumor With KRAS Mutation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-15293-002
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor
Keywords: with a KRAS mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YL-15293 (Experimental): Single arm, open, single and multiple doses; Dosage form: YL-15293 tablets Specification: 50mg, 200mg Storage conditions: refrigerated and sealed at 2-8℃
  Way of administration:
  Single-dose study: Oral administration, once a day, with warm water, fasting administration, fasting 1 hour before and 2 hours after administration. Multiple administration studies: oral administration, warm water delivery, fasting administration, fasting 1 hour before administration and 2 hours after administration, continuous administration for 21 days as a treatment cycle. The way of taking the medicine is twice a day.
  Interventions: Drug: YL-15293

INTERVENTIONS:
Drug: YL-15293 — After enrollment, patients will receive oral YL-15293 twice a day until disease progression, unacceptable adverse events, concurrent diseases prevent further study treatment, the investigator decides to withdraw the patient, the patient withdraws consent, the patient is pregnant, or for administrative reasons. After treatment, the patients will continue to be followed up for 30 days. Patients who permanently stop the study treatment for reasons other than disease progression will be followed up for disease evaluation after treatment until the start of new anti-cancer treatment, withdrawal of consent, loss of follow-up, death or until the sponsor stops the study, whichever comes first.

SUMMARY:
This is a phase 1 / 2 open label multicenter study to evaluate the maximum tolerance, safety, tolerance and PK of oral YL-15293 in patients with advanced solid tumors with KRAS mutation, so as to confirm the recommended phase 2 dose of YL-15293 and obtain the preliminary efficacy information of patients with advanced solid tumors with KRAS mutation.

DETAILED DESCRIPTION:
Dose escalation stage:

It is planned to include 21-42 subjects into 7 dose groups: 100mg/d, 200mg/d, 400mg/d, 600mg/d, 800mg/d, 1000mg/d and 1200mg/d. Three to six patients were enrolled in each dose group. 100mg/d is used as the initial dose. The dose of single administration phase is 100mg, qd, and the dose of multiple administration phase is 50mg, bid. The daily dose of the 1000mg/d dose group and above in the single administration stage is 1/2 of the daily dose, and the daily dose in the multiple administration stage is divided into two oral doses. The medication frequency (once or twice a day) and PK blood sampling point of the follow-up dose group are adjusted according to the PK parameters of the initial dose group. DLT evaluation is conducted in the first cycle (21 days).

Single-dose PK study: The drug was given once on an empty stomach in the morning on the first day, and the dose was half of the total dose of the day. Before administration (within 30 minutes before administration), pharmacokinetic samples were collected at 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours after administration. A total of 10 blood sampling points were collected, with 4ml blood taken each time .

Multi-dose PK study: 7 days after a single dose, 21 days of continuous administration is a treatment cycle, 2 times a day. On the first day, the 7th day and the 21st day, within 30 minutes before the administration, and 0.5, 1, 2, 3, 4, 6, 8, 10, 24h after the administration on the 21st day, collect the pharmacokinetics Samples, a total of 12 blood collection points, 4ml blood each time.

In addition, in the presence of DLT and SAE, a blood sample must be collected immediately for pharmacokinetic analysis.

Clinical expansion stage:

About 100-150 subjects are planned to be enrolled The sample size of NSCLC(locally advanced or metastatic G12C mutation) should be ≥ 20 cases. Select 3 or more dose groups for dose expansion,Each dose group needs about 8-50 subjects (adjusted according to the actual situation), including about 8-12 cases conduct pharmacokinetic study. The dose used for the extended test may be an incremental dose, orIt may be the intermediate dose between two incremental doses. During the study period, the researcher based on the facts response evaluation criteria in solid tumors,RECIST 1.1.

ELIGIBILITY:
Patients must meet all of the following inclusion criteria before they can be enrolled in this trial:

1. Age ≥ 18 years
2. For locally advanced or metastatic malignant solid tumors with KRAS mutations (including p.G12D, p.G12V, p.G12C, p.G12A) confirmed by histology and genomics, patients with KRAS p.G12C mutations are preferentially enrolled.

   A. For patients with NSCLC, previous first-line treatment based on platinum failed; B. For patients with colorectal cancer, at least two-line systemic treatment regimens have been experienced previously（Patients with colorectal cancer and high microsatellite instability must receive at least PD-1 or PD-L1 if clinically applicable） C. Patients with solid tumors other than NSCLC or colorectal cancer should have received systematic treatment at least once.
3. According to recist1.1 standard, there are measurable or evaluable tumor lesions
4. performance status，PS≤1
5. Estimated survival time > 3 months
6. It has a good level of organ function A. Bone marrow function needs to meet：ANC≥1.5×109/L；PLT≥100×109/L；Hb≥9g/dL B. renal function：Cr≤1.5 times the upper limit of normal value；or Creatinine clearance≥50ml/min C. liver function：total bilirubin<1.5 x ULN（For subjects with documented Gilbert syndrome,< 2.0 x ULN or subjects with indirect bilirubin levels suggesting a source of extrahepatic elevation<3.0 x ULN）；ALT and AST≤ 2.5 x ULN（If liver metastasis occurs≤ 5 x ULN） D. Coagulation function：Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper normal limit (ULN), or international normalized ratio (INR) < 1.5 or within the target range (if preventive anticoagulant therapy is performed） E). The corrected QT interval (QTcF) of Fridericia method is less than 450 ms for males and less than 470 ms for females.
7. The elution period of macromolecular drugs is ≥ 4 weeks, and that of oral fluorouracil and small molecule targeted drugs is ≥ 2 weeks
8. Fertile women must have a negative blood pregnancy test within 72 hours before receiving the first study drug;
9. For fertile men and women, they must be willing to use appropriate contraceptive methods 30 days before the first study drug administration and 120 days after the last study drug administration;
10. Did not participate in the clinical trial as a subject within 1 month before participating in the trial;
11. According to the judgment of the researcher, the compliance is high, willing to complete the test and can abide by the test scheme;
12. Voluntarily participate in this clinical trial, understand the research procedures and be able to sign the informed consent form in writing.

Exclusion criteria

Patients with any of the following items cannot be enrolled in this study:

1. Untreated patients with brain metastasis meet one or more of the following conditions：

   1. Need to use corticosteroids or dehydration treatment (except those with treated or asymptomatic brain metastases);
   2. There are significant clinical symptoms;
   3. The tumor stabilization time after radiotherapy or surgery should not exceed 4 weeks.

   (Except for patients with brain metastasis who have been treated or have no symptoms)
2. Other malignant tumors in recent five years. Basal cell carcinoma of the skin, except squamous cell carcinoma of the skin or cervical carcinoma in situ after potential treatment;
3. Myocardial infarction, symptomatic congestive heart failure (New York Heart Association > grade II), unstable angina pectoris or arrhythmia requiring drug treatment occurred within 6 months before enrollment
4. Have a history of gastrointestinal diseases or gastric surgery or inability to swallow oral drugs
5. Active infection requiring treatment
6. Patients with active hepatitis B (hepatitis B surface antigen and / or hepatitis B core antibody positive and HBV-DNA > 103 copies /mL or 200IU/mL) or hepatitis C patients (hepatitis C virus positive and / or HCV-RNA positive) or HIV positive patients are required to receive treatment.
7. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks before the first use of the study drug, or elective surgery during the trial, or therapeutic or palliative radiotherapy within 2 weeks before the first use of the study drug
8. Allergic constitution, or known history of allergy to this drug component
9. According to the researchers' judgement, there are serious diseases that may endanger the safety of patients or affect the completion of research, such as uncontrollable hypertension, uncontrollable diabetes and thyroid diseases.
10. There is fluid accumulation in the third space that cannot be controlled by drainage or other methods (such as massive identification and hydrothorax)
11. Have a clear history of neurological or mental disorders
12. The researchers believe that the subjects are not suitable to participate in this study for other reasons

In case of one or more of the following circumstances, the subject shall suspend the test:

1. Subjects asked to withdraw from the study;
2. Imaging evidence shows that the disease is progressing
3. Pregnancy events occurred during the study
4. After dose adjustment, the subject still could not tolerate the toxicity
5. The researcher considers it necessary to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) | Throughout the study for approximately 2 years
  The overall response rate (ORR) will be estimated based on the proportion of evaluable patients whose overall response (ORR) during study treatment is CR or PR. Disease response will be assessed by the investigator using RECIST v1.1.
Progression free survival, PFS | Throughout the study for approximately 2 years
  PFS, defined as the time from the first dose of study treatment to first
Overall survival, OS | Throughout the study for approximately 2 years
  The time from randomization to death for any reason
Disease control rate, DCR | Throughout the study for approximately 2 years
  The percentage of cases with remission (PR+CR) and stable lesions (SD) after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PH D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No